CLINICAL TRIAL: NCT07124819
Title: Randomized, Double-blind, Double-masked Prospective Multicenter Trial to Evaluate the Efficacy and Safety of the Oral Anticoagulant Dimolegin® Compared With Low Molecular Weight Heparin (Clexane®) as a Means of Preventing VTE in Patients Undergoing Elective Endoprosthetics of Large Joints
Brief Title: Dimolegin® (60 mg) Given Once Daily in Patients Undergoing Total Hip or Knee Replacement Compared to Enoxaparin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avexima Diol LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AVD-DIM-PН-2023-01
Record Dates: First submitted 2025-08-07; First posted 2025-08-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee; Venous Thromboembolism (VTE); Prevention
MeSH Terms: conditions — Venous Thromboembolism | interventions — enoxaparin sodium; Enoxaparin; (+-)-(1'R*,2'S*,6'R*)-(2-hydroxy-4,6-dimethoxyphenyl)(3'-methyl-2'-(3''-methylbut-2''-enyl)-6-phenylcyclohex-3'-enyl)methanone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Dimolegin® Group) (Experimental): Subgroup 1A (Hip Arthroplasty): Dimolegin® + placebo Clexane® for 35±2 days. Subgroup 1B (Knee Arthroplasty): Dimolegin® + placebo Clexane® for 14±1 days.
  Interventions: Drug: Dimolegin; Drug: Sodium enoxaparine placebo
- 2 (Clexane® Group) (Active Comparator): Subgroup 2A (Hip Arthroplasty): Clexane® + placebo Dimolegin® for 35±2 days. Subgroup 2B (Knee Arthroplasty): Clexane® + placebo Dimolegin® for 14±1 days.
  Interventions: Drug: Sodium enoxaparin; Drug: Dimolegin placebo

INTERVENTIONS:
Drug: Sodium enoxaparin — Subgroup 2A (Hip Arthroplasty): Patients undergoing total hip arthroplasty will receive Clexane® subcutaneously administered 12±1 hours before surgery starting 6-10 hours after surgery everyday for 35±2 days.
  Subgroup 2B (Knee Arthroplasty): Patients undergoing total knee arthroplasty will receive Clexane® subcutaneously administered 12±1 hours before surgery everyday for 14±1 days.
  Other Names: Clexane
  Arms: 2 (Clexane® Group)
Drug: Dimolegin — Subgroup 1A (Hip Arthroplasty): Patients undergoing total hip arthroplasty will receive Dimolegin® starting 6-10 hours after surgery everyday for 35±2 days.
  Subgroup 1B (Knee Arthroplasty): Patients undergoing total knee arthroplasty will receive Dimolegin® starting 6-10 hours after surgery everyday for 14±1 days.
  Arms: 1 (Dimolegin® Group)
Drug: Dimolegin placebo — Subgroup 2A (Hip Arthroplasty): Patients undergoing total hip arthroplasty will receive placebo Dimolegin® starting 6-10 hours after surgery everyday for 35±2 days. Subgroup 2B (Knee Arthroplasty): Patients undergoing total knee arthroplasty will receive placebo Dimolegin® starting 6-10 hours after surgery everyday for 14±1 days.
  Arms: 2 (Clexane® Group)
Drug: Sodium enoxaparine placebo — Subgroup 1A (Hip Arthroplasty): Patients undergoing total hip arthroplasty will receive palcebo Clexane® subcutaneously administered 12±1 hours before surgery starting 6-10 hours after surgery everyday for 35±2 days.
  Subgroup 2B (Knee Arthroplasty): Patients undergoing total knee arthroplasty will receive placebo Clexane® subcutaneously administered 12±1 hours before surgery everyday for 14±1 days.
  Other Names: Clexane placebo
  Arms: 1 (Dimolegin® Group)

SUMMARY:
This clinical study aims to evaluate the efficacy and safety of the anticoagulant Dimolegin® compared to low molecular weight heparin (Clexane®) for the prevention of venous thromboembolic events (VTE) in patients undergoing major joint (hip or knee) replacement surgery. The study will assess the incidence of VTE, VTE-related mortality, and all-cause mortality during different follow-up periods in both treatment groups. Additionally, the study will evaluate the frequency of bleeding events and the incidence, number, and characteristics of all adverse events associated with Dimolegin® and Clexane® therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 80.
* Patients scheduled for unilateral elective total hip or knee arthroplasty.
* The patient's voluntary informed consent.
* Negative pregnancy test result (for female patients with preserved reproductive potential).
* Patients with reproductive potential should agree to use methods of contraception according to the protocol.

Exclusion Criteria:

* Surgery for an acute fracture (<4 weeks).
* Revision or extraction arthroplasty.
* Septic arthritis.
* The only lower limb.
* Increased risk of thrombosis.
* Active bleeding or increased risk of bleeding.
* Current coagulopathy (patient's or his relative's) or congenital thrombophilia.
* Collection of at least one volume unit of donated blood (≥ 450 ml) or blood transfusion during the previous 12 weeks.
* Surgery or injury during the last 90 days.
* Diseases of the digestive system that may disrupt the absorption of the study drug.
* Significant cardiovascular diseases currently or within 6 months prior to screening.
* Active liver or biliary tract diseases.
* Creatinine clearance, calculated according to the Cockcroft-Gault formula, less than 30 ml/min.
* Positive test result for HIV, syphilis, hepatitis B and C markers.
* The development of trophic disorders of the lower extremities that are not amenable to drug treatment.
* Any condition in which, in the opinion of the researcher, surgical intervention or the use of anticoagulants is contraindicated.
* Body mass index is less than 18.5 or more than 40 kg/m2.
* Body weight for women is less than 45 kg, for men less than 57 kg and above 130 kg for both.
* Systolic blood pressure > 180 mmHg and/or diastolic blood pressure >110 mmHg.
* Hemoglobin < 105 g/l in women or < 115 g/l in men.
* Abnormal results aboratory parameters of the coagulation system (platelets, APTT, prothrombin time, INR) beyond the limits of normal values.
* An increase in ALT or ACT ≥ 2 times from the upper limit of normal (ULN) or total bilirubin ≥ 1.5 times from ULN.
* Hypersensitivity or contraindications to the administration of Dimolegin®, enoxaparin sodium, unfractionated heparin or warfarin.
* The need for constant use of parenteral or oral anticoagulants.
* The need for continuous use of antiplatelet drugs, which cannot be discontinued at least 4 days before the start of the investigational therapy.
* Systemic therapy with drugs with strong inducers and inhibitors of CYP3A4 and P-glycoprotein, which cannot be discontinued at least 7 days before the start of the investigational therapy.
* Pregnant or breast-feeding women.
* Participation in another clinical trial currently or within 90 days prior to screening.
* Affiliation to a research center, Sponsor, or contractual research organization.
* Inability to read or write; unwillingness to understand and follow the procedures of the study protocol; non-compliance with the study therapy or procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Composite endpoint i.e.: confirmed symptomatic DVT, asymptomatic DVT, non fatal PE, death of all causes | up to the follow-up visit (28±2 days after the end of therapy)

SECONDARY OUTCOMES:
Composite endpoint i.e.: confirmed symptomatic DVT, asymptomatic DVT, non fatal PE, death due to thrombosis | up to the follow-up visit (28±2 days after the end of therapy)
Switching to other anticoagulant therapy | up to the follow-up visit (28±2 days after the end of therapy)
Incidence of DVT (proximal, distal) | up to the follow-up visit (28±2 days after the end of therapy)
Incidence of non fatal PE | up to the follow-up visit (28±2 days after the end of therapy)
Incidence of symptomatic VTE | up to the follow-up visit (28±2 days after the end of therapy)
Death due to VTE | up to the follow-up visit (28±2 days after the end of therapy)
Death of all causes | up to the end of therapy (for subgroup A - up to 14±1 days, for subgroup B - up to 35±2 days)

CONTACTS AND LOCATIONS:
Locations (8):
- Russia (8):
  - Bryansk City Hospital No. 1, Bryansk
  - I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow
  - Privolzhsky Research Medical University, Nizhny Novgorod
  - Rostov State Medical University, Rostov-on-Don
  - Ryazan State Medical University named after academician I.P. Pavlov, Ryazan
  - Samara Regional Clinical Hospital named after V.D. Seredavin, Samara
  - National Research Ogarev Mordovia State University, Saransk
  - Saratov State Medical University named after V. I. Razumovsky, Saratov

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zagrekov VI, Usov AK, Vorontsov AK, Sapronova NG, Girkalo MV, Lychagin AV, Apartsin KA, Zolltukhin IA, Lomakin NV, Sychev DA. Efficacy and Safety of the Oral Anticoagulant DIMOLEGIN Compared to Enoxaparin Sodium for the Prevention of Venous Thromboembolism Following Major Joint Replacement Surgery (hip or knee arthroplasty): A Randomized, Double- Blind, Multicenter Trial. Russian Journal of Cardiology and Cardiovascular Surgery. 2025;18(5):577-585. (In Russ.). https://doi.org/10.17116/kardio202518051577